CLINICAL TRIAL: NCT00225147
Title: A Randomized, Placebo-controlled, Double Blind Phase II/III Study of the Safety and Efficacy of Recombinant Human C1 Inhibitor for the Treatment of Acute Attacks in Patients With Hereditary Angioedema
Brief Title: Recombinant Human C1 Inhibitor for the Treatment of Acute Attacks in Patients With Hereditary Angioedema
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C1 1205-01
Record Dates: First submitted 2005-09-20; First posted 2005-09-23 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Hereditary Angioedema; Angioneurotic Edema
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema | interventions — Complement C1 Inhibitor Protein; conestat alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 100 IU/kg rhC1INH (Experimental): 100 IU/kg Recombinant human C1 inhibitor
  Interventions: Drug: Recombinant Human C1 Inhibitor
- 50 IU/kg rhC1INH (Experimental): 50 IU/kg Recombinant human C1 inhibitor
  Interventions: Drug: Recombinant Human C1 Inhibitor
- Saline (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Recombinant Human C1 Inhibitor — IV
  Other Names: "rhC1INH"; Ruconest; conestat alfa
  Arms: 100 IU/kg rhC1INH; 50 IU/kg rhC1INH
Drug: placebo — saline solution
  Other Names: saline; physiological salt solution
  Arms: Saline

SUMMARY:
Hereditary angioedema ("HAE") is a genetic disorder characterized by sudden recurrent attacks of local swelling (angioedema). These attacks are often painful and disabling, and, in some cases, life-threatening. "HAE" is caused by mutations in the "C1INH" gene that lead to a decrease in the blood level of functional "C1INH". This multi-center study was designed to assess the safety and tolerability, efficacy, and pharmacokinetics/pharmacodynamics of recombinant human C1 inhibitor ("rhC1INH") in the treatment of acute hereditary angioedema attacks.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
A prospectively planned interim analysis will be performed on the double-blind data.

ELIGIBILITY:
Main Inclusion Criteria:

* Clear clinical and laboratory diagnosis of HAE
* Plasma level of functional C1INH of less than 50% of normal
* Acute abdominal, urogenital, peripheral, and/or oro-facial/pharyngeal/laryngeal HAE attack

Main Exclusion Criteria:

* Acquired angioedema
* Pregnancy or breastfeeding
* Treatment with any investigational drug within prior 30 days
* Body weight >120 kg

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2005-07; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Relan, MD, Study Director — Pharming Group N.V.
Locations (1):
- For information on sites please contact Pharming Medical Affairs Department, Leiden, Netherlands

REFERENCES:
- [Result] Zuraw B, Cicardi M, Levy RJ, Nuijens JH, Relan A, Visscher S, Haase G, Kaufman L, Hack CE. Recombinant human C1-inhibitor for the treatment of acute angioedema attacks in patients with hereditary angioedema. J Allergy Clin Immunol. 2010 Oct;126(4):821-827.e14. doi: 10.1016/j.jaci.2010.07.021. PMID 20920772
- [Derived] Bernstein JA, Relan A, Harper JR, Riedl M. Sustained response of recombinant human C1 esterase inhibitor for acute treatment of hereditary angioedema attacks. Ann Allergy Asthma Immunol. 2017 Apr;118(4):452-455. doi: 10.1016/j.anai.2017.01.029. Epub 2017 Mar 9. PMID 28284978
- [Derived] Riedl MA, Levy RJ, Suez D, Lockey RF, Baker JW, Relan A, Zuraw BL. Efficacy and safety of recombinant C1 inhibitor for the treatment of hereditary angioedema attacks: a North American open-label study. Ann Allergy Asthma Immunol. 2013 Apr;110(4):295-9. doi: 10.1016/j.anai.2013.02.007. Epub 2013 Mar 6. PMID 23535096

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the double-blind phase of the study, patients were randomized once to receive 100 IU/kg "rhC1INH", 50 IU/kg "rhC1INH" or Saline in a ratio of 1:1:1. After treatment in the double-blind phase, patients with subsequent eligible attacks could be treated with open-label 50 IU/kg "rhC1INH".
Pre-assignment Details: Patients could be enrolled into the open-label phase of the study after treatment in the double-blind phase of the study, including those enrolled but not treated in the double-blind phase.
Groups:
- 100 IU/kg "rhC1INH": Includes all subjects randomized and treated with 100 IU/kg Recombinant human C1 inhibitor in the double-blind phase
- 50 IU/kg "rhC1INH": Includes all subjects randomized and treated with 50 IU/kg Recombinant human C1 inhibitor in the double-blind phase
- Placebo: Includes all subjects randomized and treated with Placebo in the double-blind phase
- 50 IU/kg Open-label "rhC1INH": Includes all subjects treated with 50 IU/kg open-label "rhC1INH" in the open-label phase.
Period: Double-blind Phase
Arm/Group | 100 IU/kg "rhC1INH" | 50 IU/kg "rhC1INH" | Placebo | 50 IU/kg Open-label "rhC1INH"
Started | 13 | 12 | 13 | 0
Completed | 13 | 12 | 13 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Open-label Phase
Arm/Group | 100 IU/kg "rhC1INH" | 50 IU/kg "rhC1INH" | Placebo | 50 IU/kg Open-label "rhC1INH"
Started | 0 | 0 | 0 | 62
Completed | 0 | 0 | 0 | 52
Not Completed | 0 | 0 | 0 | 10
Not completed — Lost to Follow-up | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- 100 IU/kg "rhC1INH": Baseline characteristics were calculated for the modified intention to treat ("mITT") and per protocol analysis populations, which included all subjects who received 100 IU/kg "rhC1INH".
- 50 IU/kg "rhC1INH": Baseline characteristics were calculated for the modified intention to treat ("mITT") and per protocol analysis populations, which included subjects who received 50 IU/kg "rhC1INH". One (1) subject was randomized to the 50 IU/kg "rhC1INH" arm, but did not receive study drug administration and was excluded from the "mITT" analysis population.
- Placebo: Baseline characteristics were calculated for the modified intention to treat ("mITT") analysis population, which included all subjects randomized to the placebo arm.
- 50 IU/kg Open-label "rhC1INH": Baseline characteristics were calculated for the modified intention to treat ("mITT")analysis population, which included all subjects who received 50 IU/kg open-label "rhC1INH".
- Total: Total of all reporting groups
Arm/Group | 100 IU/kg "rhC1INH" | 50 IU/kg "rhC1INH" | Placebo | 50 IU/kg Open-label "rhC1INH" | Total
Number analyzed (Participants) | 13 | 12 | 13 | 39 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1 | 9 | 11
  Between 18 and 65 years | 11 | 12 | 12 | 30 | 65
  >=65 years | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 12 | 22 | 50
  Male | 5 | 4 | 1 | 17 | 27

OUTCOME MEASURES:

1. Primary Outcome: Time to Beginning of Relief of Symptoms
Description: The time to beginning of relief of symptoms at the location that showed the first visual analogue scale ("VAS") score decrease of at least 20 mm from baseline score with persistence to the next timepoint, assessment timepoints were taken on pre-scheduled time-points after study drug administration: baseline (0 minutes), 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours and 48 hours. Time to beginning of relief has been calculated as median time, by using the exact timepoints on which each assessment was performed.
Time Frame: up to 48 hours after study drug administration
Population: The full analysis set ("FAS" or "mITT") was defined as the set of patients who provided Informed Consent, were randomized and took at least one dose of the study drug administration.
Measure: Median (Full Range); unit: minutes
Groups:
- 100 IU/kg "rhC1INH": Includes all subjects enrolled and randomized to the 100 IU/kg body weight recombinant human C1 Inhibitor arm
- 50 IU/kg "rhC1INH": Includes all subjects enrolled and randomized to the 50 IU/kg body weight recombinant human C1 Inhibitor arm
- Placebo: Includes all subjects enrolled and randomized to the Saline arm
- 50 IU/kg Open-label "rhC1INH": Includes all subjects who received 50 IU/kg open-label Recombinant human C1 inhibitor
Arm/Group | 100 IU/kg "rhC1INH" | 50 IU/kg "rhC1INH" | Placebo | 50 IU/kg Open-label "rhC1INH"
Number analyzed (Participants) | 13 | 12 | 13 | 62
minutes | 68 [55 to 285] | 122 [29 to 250] | 258 [30 to 721] | 62.5 [15 to 1499]
Statistical Analysis 1: Comparison: 100 IU/kg "rhC1INH" vs Placebo; Test type: Superiority or Other; p = 0.001, Log Rank
Statistical Analysis 2: Comparison: 50 IU/kg "rhC1INH" vs Placebo; Test type: Superiority or Other; p < 0.001, Log Rank

2. Secondary Outcome: Time to Minimal Symptoms
Description: The time to minimal symptoms was the time to minimal symptoms for an attack, assessed using the Visual Analogue Scale ("VAS") score. Symptoms were said to be minimal when the "VAS" score at all locations was below 20 mm. Assessment timepoints were: baseline, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours and 48 hours. Time to minimal symtoms has been calculated by using the exact timepoints on which each assessment was performed.
Time Frame: up to 48 hours after study drug administration
Population: as for outcome 1
Measure: Median (Full Range); unit: minutes
Groups:
- 100 IU/kg "rhC1INH": Includes all subjects enrolled and randomized to the 100 IU/kg Recombinant human C1 inhibitor arm
- 50 IU/kg "rhC1INH": Includes all subjects enrolled and randomized to the 50 IU/kg Recombinant human C1 inhibitor arm
Arm/Group | 100 IU/kg "rhC1INH" | 50 IU/kg "rhC1INH" | Placebo | 50 IU/kg Open-label "rhC1INH"
Number analyzed (Participants) | 13 | 12 | 13 | 62
minutes | 245 [125 to 270] | 246.5 [243 to 484] | 1101 [970 to 1494] | 145 [124 to 256]
Statistical Analysis 1: Comparison: 100 IU/kg "rhC1INH" vs Placebo; Test type: Superiority or Other; p = 0.040, Log Rank
Statistical Analysis 2: Comparison: 50 IU/kg "rhC1INH" vs Placebo; Test type: Superiority or Other; p < 0.001, Log Rank

ADVERSE EVENTS:
Time Frame: Treatment-Emergent-Adverse-Events (TEAEs) were defined as events with start from onset of study drug administration. Serious Adverse events and Adverse events for each arm with onset dates within 7 days of study drug administration have been listed.
Groups:
- 100 IU/kg rhC1INH: Includes all subjects receiving 100 IU/kg Recombinant human C1 inhibitor
- 50 IU/kg rhC1INH: Includes all subjects receiving 50 IU/kg Recombinant human C1 inhibitor
- Placebo: Includes all subjects receiving Saline solution
- 50 IU/kg Open-label "rhC1INH": Includes all subjects receiving 50 IU/kg open-label recombinant human C1 inhibitor and subjects receiving an additional dose of 50 IU/kg "rhC1INH" within 4 hours after initial administration.
Arm/Group | 100 IU/kg rhC1INH | 50 IU/kg rhC1INH | Placebo | 50 IU/kg Open-label "rhC1INH"
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/13 | 4/62
Other Adverse Events (participants affected / at risk) | 2/13 | 2/12 | 3/13 | 18/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 IU/kg rhC1INH (N=13) | 50 IU/kg rhC1INH (N=12) | Placebo (N=13) | 50 IU/kg Open-label "rhC1INH" (N=62)
pneumonia - severe (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
vertigo - severe (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 IU/kg rhC1INH (N=13) | 50 IU/kg rhC1INH (N=12) | Placebo (N=13) | 50 IU/kg Open-label "rhC1INH" (N=62)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 12 (23)
injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vertigo (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must provide a copy of any results communication to the sponsor for review at least 30 days prior to its submission or disclosure. The sponsor may request to delete information identified by sponsor as confidential information prior to submitting such manuscript and/or abstract for publication. For a multi-center study, the investigator must wait (i) at least 24 months after the study is completed at all sites or (ii) until after the multi-center publication.